CLINICAL TRIAL: NCT01241773
Title: A Phase I, 2-panel, Open-label, Randomized, Crossover Trial in Healthy Subjects to Investigate the Pharmacokinetic Interaction Between TMC435 and Antiretroviral Agents, Efavirenz and Raltegravir, at Steady State
Brief Title: TMC435-TiDP16-C123 - A Study in Healthy Volunteers Investigating the Pharmacokinetic Interaction Between TMC435 and the Antiretroviral Agents Efavirenz and Raltegravir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR017494
Record Dates: First submitted 2010-10-21; First posted 2010-11-16 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-11

CONDITIONS: Hepatitis C Virus
Keywords: TMC435-TiDP16-C123; TMC435-C123; TMC435; HCV; Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Raltegravir Potassium; Simeprevir; efavirenz

ARMS (6):
- 001 (Experimental): TMC435 Two 75 mg capsules once daily for 14 days
  Interventions: Drug: TMC435
- 002 (Experimental): efavirenz One 600 mg tablet once daily for 14 days
  Interventions: Drug: efavirenz
- 003 (Experimental): TMC435 + efavirenz Two 75 mg TMC435 capsules + one 600 mg TMC278 tablet once daily for 14 days
  Interventions: Drug: TMC435 + efavirenz
- 004 (Experimental): TMC435 Two 75 mg capsules once daily for 7 days
  Interventions: Drug: TMC435
- 005 (Experimental): raltegravir One 400 mg tablet twice daily for 7 days
  Interventions: Drug: raltegravir
- 006 (Experimental): TMC435 + raltegravir Two 75 mg TMC435 capsules once daily and one 400 mg raltegravir tablet for 7 days
  Interventions: Drug: TMC435 + raltegravir

INTERVENTIONS:
Drug: raltegravir — One 400 mg tablet twice daily for 7 days
  Arms: 005
Drug: TMC435 + raltegravir — Two 75 mg TMC435 capsules once daily and one 400 mg raltegravir tablet for 7 days
  Arms: 006
Drug: TMC435 — Two 75 mg capsules once daily for 7 days
  Arms: 004
Drug: TMC435 + efavirenz — Two 75 mg TMC435 capsules + one 600 mg TMC278 tablet, once daily for 14 days
  Arms: 003
Drug: TMC435 — Two 75 mg capsules once daily for 14 days
  Arms: 001
Drug: efavirenz — One 600 mg tablet once daily for 14 days
  Arms: 002

SUMMARY:
The purpose of this study is to investigate the effect of steady-state concentrations of TMC435 on the steady-state pharmacokinetics of efavirenz or raltegravir , and vice versa. Steady state is a term which means that the drug has been given long enough so that the plasma concentrations will remain the same with each subsequent dose. TMC435 is being investigated for the treatment of chronic hepatitis C virus (HCV) infection. Efavirenz and raltegravir are two antiretroviral drugs for treatment of human deficiency virus (HIV) infection. Pharmacokinetics (pk) means how the drug is absorbed into the bloodstream, distributed in the body and eliminated from the body.

DETAILED DESCRIPTION:
TMC435 is being investigated for treatment of chronic hepatitis C virus (HCV) infection, in combination with Peg-IFN (pegylated interferon) and RBV (ribavirin). About 30% of all HIV infected patients are co-infected with HCV and need treatment for both infections. The results of this study will provide dosing recommendations for coadministration of TMC435 and efavirenz or raltegravir in HIV-HCV co-infected patients. This is a Phase I, open-label (both participant and investigator know the name of the medication given at certain moment), randomized (sequence of treatment with study medications is assigned by chance), crossover trial in 48 healthy volunteers to investigate the pharmacokinetic interaction between TMC435 and an antiretroviral agent (efavirenz or raltegravir), at steady state. The volunteers are being allocated to one of two panels. In Panel 1, volunteers will receive three treatments (treatment A-B-C) in a randomized order. Volunteers will receive TMC435 150 mg q.d., efavirenz 600 mg q.d. and efavirenz 600 mg q.d. + TMC435 150 mg q.d., respectively. All treatments will be administered for 14 days. There will be a washout period (a period where no study drug will be taken in view of having all the medication eliminated from the body before starting a new treatment) of at least 14 days between last intake of study medication in one session and first intake of study medication in the subsequent session. In Panel 2, volunteers will receive three treatments (treatment D-E-F) in a randomized order. Volunteers will receive TMC435 150 mg q.d., raltegravir 400 mg b.i.d. and raltegravir 400 mg b.i.d. + TMC435 150 mg q.d., respectively. All treatments will be administered for 7 days. There will be a washout period of at least 7 days. Pharmacokinetic profiles of all three compounds will be determined through blood samples taken at regular intervals during the study. Safety and tolerability will be assessed during the study period and in follow-up. Blood and urine samples, electrocardiogram (ECG) and vital signs (blood pressure and heart rate) will be taken at screening, before medication intake on Days 1 and 14 and on Day 15 in each session of Panel 1, before medication intake on Days 1 and 7 and on Day8 in each session of Panel 2, 6 hours post dose on Day14 and Day7 in Panel 1 and 2, respectively and at the 2 follow up visits at 1 week and 4-5 weeks after last dose of study medication in the last session. A physical examination will be performed at screening, on Day-1 (= day before first medication intake in each session for both panels) and on Day15 in Panel 1, on Day-1 and on Day8 of Panel 2 and during the 2 follow up visits. Each volunteer will receive 3 treatments for 14 or 7 days (Panel 1 and 2, respectively), minimum 14 or 7 days apart from each other (Panel 1 and 2, respectively). Volunteers in Panel 1 will take oral TMC435 150 mg q.d., oral efavirenz 600 mg q.d. and combined. Volunteers in Panel 2 will take oral TMC435 150 mg q.d., oral raltegravir 400 mg b.i.d. and combined.

ELIGIBILITY:
Inclusion Criteria:

* No-smoker for at least 3 months
* Body Mass Index of 18.0 to 30.0 kg/m2
* Healthy based on a medical evaluation including medical history, physical examination, blood tests and electrocardiogram

Exclusion Criteria:

* Infection with Hepatitis A, B or C Virus
* Infection with the Human Immunodeficiency Virus (HIV)
* History of, or any current medical condition which could impact the safety of the participant in the study
* Having previously participated in a multiple-dose trial with TMC435
* Having previously participated in more than 3 single-dose trials with TMC435.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Absorption of TMC435 following co-administration with efavirenz, and vice versa. | Measured on Day1, 12, 13, 14, 15, 16, 17 and 18 for both drugs in eaach treatment in Panel 1.
Absorption of TMC435 following co-administration with raltegravir, and vice versa. | Measured on Day1, 5, 6, and 7 for both drugs in each treatment of Panel2 and on Day8-11 for TMC435 only in treatment D and F in Panel 2.

SECONDARY OUTCOMES:
Number of participants with Adverse Events as a measure of Safety and Tolerability - TMC435 and efavirenz. | 98 to 103 days (till and including last safety follow-up visit) for Panel 1
Number of participants with Adverse Events as a measure of Safety and Tolerability - TMC435 and raltegravir. | 63 to 68 days (till and including last safety follow-up visit) for Panel 2

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited
Locations (1):
- Berlin, Germany